CLINICAL TRIAL: NCT06319586
Title: The Radial Forearm Flap In Reconstruction Of Upper Limb Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelmawla Mohamed, Resident of Orthopaedic department, Sohag University Hospitals, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-02-08MS
Record Dates: First submitted 2024-03-10; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: for Upper Limb Soft Tissue Coverage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radial Forearm Flap — * Elevate the flap from ulnar to radial side toward the FCR
  * Elevate flap from radial to ulnar side to the brachioradialis tendon. Ligate and divide the radial artery and venae comitantes distally.
  * incise the skin over the cephalic vein proximally to the cubital fossa. Identify the venous branching pattern and perforating vein.
  * Elevate the skin and subcutaneous paddles proximally off of the FCR and brachioradialis.
  * Define the venous anatomy at the cubital fossa. In most cases, the median basilic vein and continuation of the median vein contribution to the cephalic vein can be harvested proximal to the perforating vein. This anatomy allows two large veins to be harvested that drain both the deep and superficial systems. Occasionally, one large vein will be identified.
  * Closure is performed by harvesting a 0.018-inch skin graft to cover the donor defect. The radial skin edge should be advanced to cover the exposed radial nerve.

SUMMARY:
The radial forearm flap is a very useful and versatile flap with a long vascular pedicle and a thin, pliable skin. It's used in reconstruction of the mutilated hand as a reverse pedicled flap. The dominant pedicle is the radial artery, with venous outflow through the dual system of the venae comitantes and cephalic vein. Sensory innervation may be derived from the medial and lateral antebrachial cutaneous nerves. The radial forearm flap offers the advantage of a large area of donor tissue from the involved extremity with the potential for inclusion of bone, nerve, and tendon grafts. Sacrifice of the radial artery has not been associated with significant patient symptoms However, the donor defect can be troublesome, frequently requiring skin grafting directly over the paratenon of the flexor tendons, producing an undesirable donor site appearance

ELIGIBILITY:
Inclusion Criteria:

* patients aging 5 to 80 years.
* Soft Tissue defects following MCA injuries.
* Defect size less than 30 cm

Exclusion Criteria:

* Peripheral vascular disease
* Underling bone osteomyelitis
* Unhealthy skin of volatile aspect of donor forearm
* Defect more than 30 cm
* Ulnar artery previous ligated

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Viability of the flap | 12 months
  viability of the flap including color, warmth, capillary refill, smell and turgor

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noaman HH. Management of upper limb bone defects using free vascularized osteoseptocutaneous fibular bone graft. Ann Plast Surg. 2013 Nov;71(5):503-9. doi: 10.1097/SAP.0b013e3182a1aff0. PMID 24126338
- [Background] Noaman HH, Shiha AE. Repeated upper limb salvage in a case of severe traumatic soft-tissue and brachial artery defect. Microsurgery. 2002;22(6):249-53. doi: 10.1002/micr.10045. PMID 12375291
- [Background] Noaman HH. Salvage of complete degloved digits with reversed vascularized pedicled forearm flap: a new technique. J Hand Surg Am. 2012 Apr;37(4):832-6. doi: 10.1016/j.jhsa.2012.01.032. Epub 2012 Mar 6. PMID 22397844
- [Background] Kaufman MR, Jones NF. The reverse radial forearm flap for soft tissue reconstruction of the wrist and hand. Tech Hand Up Extrem Surg. 2005 Mar;9(1):47-51. doi: 10.1097/01.bth.0000154479.20226.22. PMID 16092819